CLINICAL TRIAL: NCT01939496
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Blood Pressure Reduction With Ambulatory Blood Pressure Monitoring (ABPM), Safety, and Tolerability of Canagliflozin in the Treatment of Subjects With Hypertension and Type 2 Diabetes Mellitus
Brief Title: Evaluation of Blood Pressure Reduction, Safety, and Tolerability of Canagliflozin in Patients With Hypertension and Type 2 Diabetes Mellitus on Stable Doses of Anti-hyperglycemic and Anti-hypertensive Agents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR102208; 28431754DIA4002 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: Diabetes Mellitus, Type 2; Hypertension; Canagliflozin; JNJ 28431754; Sodium-Glucose Transporter 2; Blood Glucose; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Canagliflozin 100 mg (Experimental): Each patient will receive 100 mg of canagliflozin once daily for 6 weeks.
  Interventions: Drug: Canagliflozin
- Canagliflozin 300 mg (Experimental): Each patient will receive 300 mg of canagliflozin once daily for 6 weeks.
  Interventions: Drug: Canagliflozin
- Placebo (Placebo Comparator): Each patient will receive matching placebo once daily for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin — One 100 mg or 300 mg over-encapsulated tablet orally (by mouth) in addition to the patient's anti-hyperglycemic agents (AHA) regimen used in accordance with local prescribing information.
  Arms: Canagliflozin 100 mg; Canagliflozin 300 mg
Drug: Placebo — One matching placebo capsule orally in addition to the patient's anti-hyperglycemic agents (AHA) regimen used in accordance with local prescribing information.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of canagliflozin (JNJ-28431754) on blood pressure reduction, compared to placebo, in patients with hypertension and type 2 diabetes mellitus and who are on stable doses of anti-hyperglycemic and anti-hypertensive agents. Overall safety and tolerability of canagliflozin will be assessed.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double blind (neither the patient nor the study doctor will know the name of the assigned treatment), parallel-group, 3-arm (patients will be assigned to 1 of 3 treatment groups) multicenter study to determine the effect of canagliflozin (100 mg and 300 mg) on blood pressure (BP) reduction compared to placebo (a pill that looks like all the other treatments but has no real medicine) in patients with hypertension and type 2 diabetes mellitus (T2DM). The study will consist of 3 phases: a screening phase, a double-blind treatment phase and a follow-up period. Approximately 153 participants will be randomly assigned to 1 of 3 treatment groups (in a 1:1:1 ratio) in the double-blind treatment phase to receive canagliflozin 100 mg, canagliflozin 300 mg or placebo for 6 weeks. The total duration of participation in this study will be approximately 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of type 2 diabetes mellitus
* patients with hypertension (seated office SBP of >=130 mmHg and <160 mmHg and seated office DBP of >= 70 mmHg at screening and at Week -2
* patients on stable doses of 1 to 3 anti-hypertensive agents for at least 5 weeks before screening
* patients on stable doses of 1 to 3 oral anti-hyperglycemic agents which must include metformin, for at least 8 weeks before screening

Exclusion Criteria:

* a history of diabetic ketoacidosis
* type 1 diabetes mellitus (T1DM)
* pancreas or beta-cell transplantation
* fasting C-peptide <0.70 ng/mL (0.23 nmol/L)
* body mass index <30 kg/m2
* has ongoing, inadequately controlled thyroid disorder
* has a history of cardio-renal disease that required treatment with immunosuppressive therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (57):
- United States (54):
  - Birmingham, Alabama
  - Gulf Shores, Alabama
  - Avondale, Arizona
  - Phoenix, Arizona
  - Glendale, California
  - Los Angeles, California
  - Newport Beach, California
  - Pismo Beach, California
  - Rancho Cucamonga, California
  - Roseville, California
  - Sacramento, California
  - Spring Valley, California
  - Tustin, California
  - Denver, Colorado
  - Brandon, Florida
  - Doral, Florida
  - Fort Lauderdale, Florida
  - Lake Worth, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - West Palm Beach, Florida
  - Perry, Georgia
  - Rincon, Georgia
  - Indianapolis, Indiana
  - Topeka, Kansas
  - Lexington, Kentucky
  - Mandeville, Louisiana
  - Marrero, Louisiana
  - Metairie, Louisiana
  - Auburn, Maine
  - Elkridge, Maryland
  - Dearborn, Michigan
  - Kalamazoo, Michigan
  - Jackson, Mississippi
  - St Louis, Missouri
  - Morganville, New Jersey
  - Whiting, New Jersey
  - Albuquerque, New Mexico
  - Raleigh, North Carolina
  - Oklahoma City, Oklahoma
  - Altoona, Pennsylvania
  - Jenkintown, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Plano, Texas
  - Sugar Land, Texas
  - Salt Lake City, Utah
  - Renton, Washington
- Puerto Rico (3):
  - Carolina
  - Ponce Pr
  - Trujillo Alto

REFERENCES:
- [Derived] Pfeifer M, Townsend RR, Davies MJ, Vijapurkar U, Ren J. Effects of canagliflozin, a sodium glucose co-transporter 2 inhibitor, on blood pressure and markers of arterial stiffness in patients with type 2 diabetes mellitus: a post hoc analysis. Cardiovasc Diabetol. 2017 Feb 27;16(1):29. doi: 10.1186/s12933-017-0511-0. PMID 28241822

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 504 participants were screened. Of which, 171 participants were randomized to study treatment. 2 participants were randomized but not dosed.
Groups:
- Placebo: Participants were received matching placebo overencapsulated tablets orally once daily for 6 Weeks.
- Canagliflozin 100 Milligram (mg): Participants were received Canagliflozin 100 mg overencapsulated tablets orally once daily for 6 Weeks.
- Canagliflozin 300 mg: Participants were received Canagliflozin 300 mg overencapsulated tablets orally once daily for 6 Weeks.
Period: Overall Study
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Started | 56 | 57 | 56
Completed | 47 | 54 | 54
Not Completed | 9 | 3 | 2
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Blood Pressure Withdrawal Criteria | 0 | 1 | 0
Not completed — Other | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants who took at least 1 dose of double blind study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Total
Number analyzed (Participants) | 56 | 57 | 56 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 46 | 45 | 129
  >=65 years | 18 | 11 | 11 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (9.52) | 57.8 (8.74) | 58.3 (6.88) | 58.6 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 25 | 71
  Male | 33 | 34 | 31 | 98

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean 24-Hour Systolic Blood Pressure (SBP) to Week 6
Description: The blood pressure (BP) was evaluated by Ambulatory Blood Pressure Monitoring (ABPM) for all participants based on the 24-hour BP recordings.
Time Frame: Baseline and Week 6
Population: The full analysis set included all randomized participants who took at least 1 dose of double blind study medication. Here, "n" specifies those participants who were evaluated for this outcome measure at given time point. Missing data was imputed using last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
millimeter of mercury (mmHg)
  Baseline (n=56,57,56) | 136.7 (10.293) | 136.5 (11.501) | 139.6 (10.925)
  Change From Baseline at Week 6 (n=54,54,55) | -1.26 (9.864) | -4.78 (8.327) | -7.31 (11.409)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 Milligram (mg); Test type: Superiority or Other; p = 0.062, ANCOVA; Difference of Least Square Means = -3.29, 95% CI 2-sided [-6.743 to 0.163], Standard Error of Mean 1.748
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.006, ANCOVA; Difference of Least Square Means = -4.93, 95% CI 2-sided [-8.382 to -1.469], Standard Error of Mean 1.750

2. Secondary Outcome: Change From Baseline in Mean 24-Hour Systolic Blood Pressure (SBP) to Day 2
Description: as for outcome 1
Time Frame: Baseline and Day 2
Population: The full analysis set included all randomized participants who took at least 1 dose of double blind study medication. Here, "n" specifies those participants who were evaluated for this outcome measure at given time point. Missing data was imputed using LOCF method.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
millimeter of mercury (mmHg)
  Baseline (n=56,57,56) | 136.7 (10.293) | 136.5 (11.501) | 139.6 (10.925)
  Change From Baseline at Day 2 (n=50,50,50) | 0.49 (8.592) | -1.78 (6.924) | -1.97 (7.343)

3. Secondary Outcome: Change From Baseline in the Mean 24-Hour Diastolic Blood Pressure (DBP) to Day 2 and to Week 6
Description: as for outcome 1
Time Frame: Baseline, Day 2 and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
millimeter of mercury (mmHg)
  Baseline (n=56,57,56) | 78.36 (7.330) | 78.01 (8.093) | 79.31 (7.899)
  Change From Baseline at Day 2 (n=50,50,50) | 1.01 (5.197) | -0.85 (4.155) | -0.45 (4.540)
  Change From Baseline at Week 6 (n=54,54,55) | -0.26 (5.345) | -2.18 (4.870) | -3.27 (6.462)

4. Secondary Outcome: Change From Baseline in Mean Daytime Systolic Blood Pressure (SBP) to Day 2 and to Week 6
Description: The diurnal rise (daytime) in blood pressure (BP) was evaluated by Ambulatory Blood Pressure Monitoring (ABPM) for all participants based on the 24-hour BP recordings.
Time Frame: Baseline, Day 2 and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
millimeter of mercury (mmHg)
  Baseline (n=56,57,56) | 139.4 (10.343) | 139.6 (11.295) | 142.8 (11.435)
  Change From Baseline at Day 2 (n=50,50,50) | 0.96 (9.494) | -2.06 (7.309) | -1.16 (7.579)
  Change From Baseline at Week 6 (n=54,54,55) | -0.65 (9.874) | -5.05 (8.656) | -7.36 (11.660)

5. Secondary Outcome: Change From Baseline in Mean Daytime Diastolic Blood Pressure (DBP) to Day 2 and to Week 6
Description: as for outcome 4
Time Frame: Baseline, Day 2 and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
millimeter of mercury (mmHg)
  Baseline (n=56,57,56) | 80.84 (7.656) | 80.53 (8.252) | 81.81 (8.377)
  Change From Baseline at Day 2 (n=50,50,50) | 1.21 (5.579) | -1.08 (4.519) | 0.03 (4.772)
  Change From Baseline at Week 6 (n=54,54,55) | -0.20 (5.257) | -2.39 (5.413) | -3.23 (6.557)

6. Secondary Outcome: Change From Baseline in Mean Nighttime Systolic Blood Pressure (SBP) to Day 2 and to Week 6
Description: The nocturnal fall (nighttime) in blood pressure (BP) was evaluated by Ambulatory Blood Pressure Monitoring (ABPM) for all participants based on the 24-hour BP recordings.
Time Frame: Baseline, Day 2 and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
millimeter of mercury (mmHg)
  Baseline (n=56,57,56) | 129.3 (12.128) | 128.3 (14.527) | 130.2 (12.727)
  Change From Baseline at Day 2 (n=50,50,50) | -0.19 (8.801) | -1.02 (8.723) | -4.37 (10.682)
  Change From Baseline at Week 6 (n=54,54,55) | -3.49 (12.469) | -4.33 (11.506) | -6.98 (12.880)

7. Secondary Outcome: Change From Baseline in Mean Nighttime Diastolic Blood Pressure (DBP) to Day 2 and to Week 6
Description: as for outcome 6
Time Frame: Baseline, Day 2 and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
millimeter of mercury (mmHg)
  Baseline (n=56,57,56) | 71.57 (8.100) | 71.10 (9.091) | 72.31 (8.515)
  Change From Baseline at Day 2 (n=50,50,50) | 0.87 (6.282) | -0.23 (5.764) | -2.24 (6.037)
  Change From Baseline at Week 6 (n=54,54,55) | -0.98 (7.749) | -1.73 (6.475) | -3.42 (8.056)

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) to Week 6
Description: The fasting plasma glucose was evaluated.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
millimoles per liter (mmol/L)
  Baseline (n=56,57,56) | 9.84 (2.435) | 9.69 (2.085) | 9.38 (2.000)
  Change From Baseline at Week 6 (n=55,54,55) | -0.38 (2.727) | -0.03 (2.702) | -1.27 (2.164)

9. Secondary Outcome: Change From Baseline in Body Weight to Week 6
Description: Body weight was evaluated.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
Kilogram (kg)
  Baseline (n=56,57,56) | 91.65 (17.525) | 95.32 (22.201) | 96.06 (20.227)
  Change From Baseline at Week 6 (n=54,55,56) | 0.14 (2.326) | -0.98 (1.964) | -1.47 (2.160)

10. Secondary Outcome: Change From Baseline in Seated Office Blood Pressure (BP) to Day 2, to Week 3, and to Week 6
Description: The seated office blood pressure (BP) was evaluated for all participants based on the 24-hour BP recordings. SBP=Systolic Blood Pressure and DBP=Diastolic Blood Pressure.
Time Frame: Baseline, Day 2, Week 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
millimeter of mercury (mmHg)
  SBP: Baseline (n=56,57,56) | 137.7 (8.581) | 138.5 (11.102) | 139.2 (8.832)
  SBP: Change From Baseline at Day 2 (n=55,57,56) | -3.24 (10.045) | -2.06 (8.971) | -5.11 (8.768)
  SBP: Change From Baseline at Week 3 (n=55,57,56) | -5.95 (10.373) | -7.53 (10.825) | -10.6 (11.340)
  SBP: Change From Baseline at Week 6 (n=55,57,56) | -3.36 (13.807) | -4.98 (11.430) | -7.38 (16.248)
  DBP: Baseline (n=55,57,56) | 82.67 (8.571) | 82.37 (7.673) | 83.02 (8.155)
  DBP: Change From Baseline at Day 2 (n=55,57,56) | -2.61 (6.259) | -0.26 (6.217) | -0.87 (5.688)
  DBP: Change From Baseline at Week 3 (n=55,57,56) | -2.84 (6.664) | -2.22 (6.226) | -4.23 (6.267)
  DBP: Change From Baseline at Week 6 (n=55,57,56) | -1.78 (9.271) | -1.52 (6.652) | -2.43 (7.479)

11. Secondary Outcome: Change From Baseline in Standing Office Blood Pressure (BP) to Day 2, to Week 3, and to Week 6
Description: The standing office blood pressure (BP) was evaluated for all participants based on the 24-hour BP recordings. SBP=Systolic Blood Pressure and DBP=Diastolic Blood Pressure.
Time Frame: Baseline, Day 2, Week 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
millimeter of mercury (mmHg)
  SBP: Baseline (n=56,57,56) | 140.3 (10.067) | 139.3 (11.801) | 140.8 (9.058)
  SBP: Change From Baseline at Day 2 (n=55,57,56) | -4.36 (10.293) | -2.46 (12.133) | -5.91 (11.617)
  SBP: Change From Baseline at Week 3 (n=55,57,56) | -6.55 (13.178) | -7.12 (12.503) | -11.9 (14.226)
  SBP: Change From Baseline at Week 6 (n=55,57,56) | -3.76 (17.651) | -7.95 (13.722) | -11.3 (16.872)
  DBP: Baseline (n=55,57,56) | 85.79 (8.608) | 85.25 (8.354) | 86.09 (7.349)
  DBP: Change From Baseline at Day 2 (n=55,57,56) | -0.65 (8.945) | -0.60 (8.914) | -1.32 (7.515)
  DBP: Change From Baseline at Week 3 (n=55,57,56) | -2.91 (8.341) | -3.47 (7.117) | -5.36 (6.632)
  DBP: Change From Baseline at Week 6 (n=55,57,56) | -0.89 (9.875) | -2.51 (7.280) | -4.55 (8.052)

12. Secondary Outcome: Change From Baseline in Seated Heart Rate (HR) to Day 2, to Week 3, and to Week 6
Description: The seated heart rate was evaluated.
Time Frame: Baseline, Day 2, Week 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
beats per minute
  Baseline (n=56,57,56) | 79.57 (14.597) | 75.05 (8.574) | 78.13 (11.060)
  Change From Baseline at Day 2 (n=55,57,56) | -1.40 (15.412) | 3.05 (7.909) | 1.68 (9.219)
  Change From Baseline at Week 3 (n=55,57,56) | -2.24 (15.412) | 1.70 (7.305) | -0.89 (8.800)
  Change From Baseline at Week 6 (n=55,57,56) | -2.24 (14.004) | 1.07 (8.351) | -1.16 (8.083)

13. Secondary Outcome: Change From Baseline in Standing Heart Rate (HR) to Day 2, to Week 3, and to Week 6
Description: The standing heart rate was evaluated.
Time Frame: Baseline, Day 2, Week 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
beats per minute
  Baseline (n=56,57,56) | 82.54 (8.826) | 78.65 (9.259) | 81.86 (11.949)
  Change From Baseline at Day 2 (n=55,57,56) | 0.27 (8.350) | 4.32 (8.403) | 2.79 (9.689)
  Change From Baseline at Week 3 (n=55,57,56) | -0.89 (10.322) | 3.47 (9.383) | 0.48 (9.217)
  Change From Baseline at Week 6 (n=55,57,56) | -0.07 (9.465) | 1.44 (9.200) | -0.68 (8.547)

14. Secondary Outcome: Change From Baseline in the Difference in Seated Office Blood Pressure (BP) and Standing Office BP to Day 2, to Week 3, and to Week 6
Description: The difference in seated office blood pressure and standing office blood pressure was evaluated.
Time Frame: Baseline, Day 2, Week 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
millimeter of mercury (mmHg)
  Baseline (n=56,57,56) | 2.65 (7.914) | 0.78 (8.964) | 1.55 (8.231)
  Change From Baseline at Day 2 (n=55,57,56) | -1.13 (10.991) | -0.39 (11.097) | -0.80 (9.078)
  Change From Baseline at Week 3 (n=55,57,56) | -0.60 (10.921) | 0.40 (8.562) | -1.27 (9.873)
  Change From Baseline at Week 6 (n=55,57,56) | -0.41 (11.875) | -2.96 (8.397) | -3.90 (11.566)

15. Secondary Outcome: Change From Baseline in the Difference in Seated Heart Rate (HR) and Standing HR to Day 2, to Week 3, and to Week 6
Description: The difference in seated heart rate and standing heart rate was evaluated.
Time Frame: Baseline, Day 2, Week 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 57 | 56
beats per minute
  Baseline (n=56,57,56) | 2.96 (14.752) | 3.60 (5.168) | 3.73 (4.232)
  Change From Baseline at Day 2 (n=55,57,56) | 1.67 (14.562) | 1.26 (6.802) | 1.11 (5.786)
  Change From Baseline at Week 3 (n=55,57,56) | 1.35 (16.008) | 1.77 (6.538) | 1.38 (5.262)
  Change From Baseline at Week 6 (n=55,57,56) | 2.16 (15.975) | 0.37 (7.203) | 0.48 (4.472)

ADVERSE EVENTS:
Time Frame: Screening up to post-treatment Phase (30 days after the last dose of study medication)
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Serious Adverse Events (participants affected / at risk) | 1/56 | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 1/56 | 4/57 | 3/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | Canagliflozin 100 Milligram (mg) (N=57) | Canagliflozin 300 mg (N=56)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | Canagliflozin 100 Milligram (mg) (N=57) | Canagliflozin 300 mg (N=56)
Nasopharyngitis (Infections and infestations) | 0 | 3 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.